CLINICAL TRIAL: NCT04583449
Title: Mental Imagery to Increase Face Covering Use in UK-based Public Places During the COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East London (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Principal Investigator, Dominic Conroy, Principal Investigator, University of East London
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: ETH2021-0006
Record Dates: First submitted 2020-10-02; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Viral Infection; Covid19
MeSH Terms: conditions — Virus Diseases; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Outcome imagery (Experimental): Outcome imagery condition participants will be asked to visualize themselves successfully wearing a face covering in all required public places/situations over coming week, and to imagine how they would feel. The importance of imagining distinctive relevant visual imagery linked to having successfully routinely worn face covering will be underscored in this passage. Outcome imagery participants will then be asked to write in a free-text box how they would feel having successfully worn a face covering in required public places/situations over the week ahead.
  Interventions: Behavioral: Mental imagery
- Process imagery (Experimental): Process imagery condition participants will be asked to visualize the kinds of strategies involved in successfully wearing a face covering in all required public places/situations over the coming week. The importance of imagining distinctive relevant visual imagery linked to having effective strategies involved in successfully wearing a face covering in required public places/situations over the week ahead will be underscored in this passage. Process imagery participants will then be asked to write in a free-text box about the kinds of strategies that would be involved in successfully wearing a face covering in all required public places/situations over the coming week.
  Interventions: Behavioral: Mental imagery
- Combined imagery (outcome imagery and process imagery) (Experimental): A third experimental condition will receive both outcome and process imagery exercises to read and complete in sequential order.
  Interventions: Behavioral: Mental imagery
- Public health message (No Intervention): A fourth condition will involve viewing a UK Government public health message (HM Government, 2020) circulated on social media as an image concerning the importance of wearing face covering while in public places.

INTERVENTIONS:
Behavioral: Mental imagery — Mental imagery involves the mental representation of a future event, action, or task. By imitating or rehearsing this mental event or series of events" (Taylor et al., 1998, p. 430) mental imagery interventionists theorise that an individual's preparation for, and motivation toward, a future action can be made more likely. Mental imagery involves an individual following a set of pre-defined exercises involving thinking about, visualising and writing about a health-related action. Mental imagery exercises can involve focusing on anticipated positive/beneficial outcomes of an action (outcome imagery) or imagery relating to the anticipated strategies/preparation that would be required to successfully execute a pre-defined action (process imagery).
  Arms: Combined imagery (outcome imagery and process imagery); Outcome imagery; Process imagery

SUMMARY:
Wearing face coverings in enclosed public spaces is a key public health measure to limit viral spread during the 2020 Covid-19 pandemic. Health psychologists are interested in developing interventions that can increase the likelihood of health-adherent and protective behaviours being consistently undertaken at a general population level. Mental imagery interventions are one way in which behavioural scientists and health psychologists try to encourage behaviour change. Mental imagery involves thinking about, and then writing about, anticipated positive outcomes or key practical requirements of a defined health-related action (e.g. 'moderate alcohol consumption'; 'engaging in regular physical activity'). For this project, the investigators are exploring a mental imagery intervention created to encourage regular and consistent wearing of face coverings in public places where this is currently required in the UK. The investigators will test whether engaging in a mental imagery exercise results in any improvement in wearing a face covering (or intention to wear a face covering) one month later relative to reading a public health message about face coverings. In addition, the investigators will explore belief-based and personality-related factors that might make a difference to the effectiveness of the mental imagery intervention.

DETAILED DESCRIPTION:
Background The 2020 Covid-19 pandemic has required wide-ranging efforts to minimize the spread of the virus and to protect those most vulnerable to becoming unwell as a result of viral infection. These measures include social distancing, regular hand washing and wearing face coverings in public places where an individual is, inevitably, in closer proximity to non-household others than when not in a public place.

The evidence base for using face coverings in the context of the Covid-19 virus has been mixed and is applied in different ways in different countries. However, there is scientific consensus has been that wearing a face covering is likely to decrease viral transmissibility and, relatedly, substantially reduce the death toll and economic impact of the pandemic. The scientific evidence suggests that face coverings primarily offer protection to other people from the person wearing the face covering (who may, knowingly or not, been infected with the virus) rather than offering the person wearing the face covering personal protection themselves. In the UK, the most recent government advice (at time of writing, published on 7th August 2020) supports the use of face coverings.

Previous studies have suggested that varied demographic and belief-based factors (including perceived benefits) may influence variation in individuals' willingness to wear a face covering in the context of a viral epidemic/pandemic past and present. The Covid-19 pandemic is particular in the sense that the risk of viral infection is understood to be greatest to individuals other than the wearer of the face covering and, for this reason, psychological theories concerned with risk susceptibility/vulnerability (e.g. Protection Motivation Theory; Health Belief Model) may have less predictive utility in the context of the 2020 pandemic. However, other social-cognitive psychological theory may offer valuable insights into factors linked to face covering adherence. For example, variation in face covering wearing adherence would be predicted by traditional behavioural science theory as closely linked to a range of key beliefs about the target behaviour. Relevant belief-related factors include attitudes towards face covering (i.e. whether an individual holds (un)favourable beliefs about face covering are held), subjective norms towards face covering (e.g. whether an individual believes that important others such as friends and family hold (un)favourable beliefs about face covering), and perceived behavioural control towards face covering (i.e. the extent to which an individual believes they possess control over deciding to wear a face covering). Whether an individual believes they possess a high level of skill in using face coverings in required situations (i.e. public places/spaces) would also be theorized to predict face covering behaviour.

A further consideration linked to individual adherence to face covering requirements is what 'type' of person that individual is in terms of various relevant personality traits. For example, a relatively conscientious person might be expected to be more likely to routinely wear a face covering to protect individuals in close proximity from the risk of viral infection. Similarly, face covering adherence might be more likely among individuals whose personalities are characterised by humanistic, beneficent orientations towards other people. By contrast, an individual who self-reports high levels of narcissism, may be less likely to wear a face covering given that wearing a face covering might clash with their relatively vain/egotistical self-image.

In summary, this study aims to determine if different types of mental imagery intervention impact on face covering intentions and face covering adherence at a follow-up time point. The second study aim is to explore, through exploratory analyses, whether individual differences in light triad traits, conscientiousness, and narcissism will influence the impact of imagery interventions. Thirdly, the moderating role of social-cognitive variables of intervention effects will be explored. Fourthly, variation in 'imagery ability' (how capable individuals are at visualizing future actions) will be examined as a mediator of potential intervention effects.

Research questions

1. Do mental imagery exercises increase intentions to use face coverings in public where required?
2. Do mental imagery exercises increase self-reported wearing of face coverings in public where required?
3. Do light triad personality traits moderate the relationship between condition allocation (imagery or not) and self-reported face covering wearing intention or action?
4. Do Theory of Planned Behaviour variables moderate/mediate the relationship between condition allocation (imagery or not) and self-reported face covering wearing intention or action?
5. Does imagery ability moderate/mediate the relationship between condition allocation (imagery or not) and self-reported face covering wearing intention or action?

Hypotheses

It is hypothesised that individuals assigned to any imagery intervention condition will report:

1. Significantly higher intentions to wear face coverings in public places where these are required, relative to the control condition at T2 (primary outcome; hypothesis 1).
2. Significantly higher levels of self-reported face covering relative to the control condition at T3 (primary outcome; hypothesis 2).
3. Significantly more favourable attitudes, subjective norms, barrier self-efficacy and perceived behavioural control linked to face covering wearing at T2 and T3 (hypotheses 3 and 4).
4. Finally, it is hypothesied that imagery intervention effects on primary outcome variables at T2 and T3 will be conditional on being more conscientious, less narcissistic, and being characterised by higher levels of 'light triad' personality traits (hypothesis 5).

ELIGIBILITY:
Inclusion Criteria:

* 18+ year old adults

Exclusion Criteria:

* Not currently living in the UK

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Face covering wearing consistency | 4 weeks post-intervention
  Self-reported single item response statement with a Likert-type response. Minimum value = 1; maximum value = 5 (a higher score indicates a better outcome).
Face covering wearing intention | 4 weeks post-intervention
  Self-reported three item response scale with Likert-type responses. Minimum value = 1; maximum value = 5 (a higher score indicates a better outcome).

SECONDARY OUTCOMES:
Attitude toward wearing a face covering | 4 weeks post-intervention
  Self-reported 3 item response scale with Likert-type responses. Minimum value = 1; maximum value = 5 (a higher score indicates a worse outcome).
Injunctive norm beliefs about wearing a face covering | 4 weeks post-intervention
  Self-reported 2 item response scale with Likert-type responses. Minimum value = 1; maximum value = 5 (a higher score indicates a better outcome).
Descriptive norm beliefs about wearing a face covering | 4 weeks post-intervention
  Self-reported 2 item response scale with Likert-type responses. Minimum value = 1; maximum value = 5 (a higher score indicates a better outcome).
Perceived behavioural control over wearing a face covering | 4 weeks post-intervention
  Self-reported 3 item response scale with Likert-type responses. Minimum value = 1; maximum value = 5 (a higher score indicates a better outcome).
Barrier self-efficacy to wearing a face covering | 4 weeks post-intervention
  Self-reported 6 item response scale with Likert-type responses. Minimum value = 1; maximum value = 5 (a higher score indicates a better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- University of East London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We will share the anonymised data as a Supplementary file when submitting a research write-up as an article to a suitable academic journal.
Supporting Information: Study Protocol
Time Frame: Data will be made available on completion of article publication. Data will be made permanently available.

REFERENCES:
- [Derived] Conroy D. Mental imagery interventions to promote face covering use among UK university students and employees during the COVID-19 pandemic: study protocol for a randomized controlled trial. Trials. 2022 Jan 18;23(1):51. doi: 10.1186/s13063-021-05852-y. PMID 35042564